CLINICAL TRIAL: NCT00251355
Title: A Phase I Study of Gemcitabine, 5-Fluorouracil, and Radiation Therapy in the Treatment of Locally Unresectable Non-Metastatic Pancreatic Cancer
Brief Title: Gemcitabine, 5-Fluorouracil, and Radiation Therapy in the Treatment of Non-Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Charles S. Fuchs, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-105
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Pancreatic Cancer
Keywords: gemcitabine; 5-fluorouracil; 5-FU; unresectable pancreatic cancer; non-metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 5-FU/gemcitabine/RT (Experimental)
  Interventions: Drug: Gemcitabine; Drug: 5-Fluorouracil; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine, IV bolus administered weekly (weeks 1-6) at least 4 hours before that day's radiation therapy.
Drug: 5-Fluorouracil — 5-FU via continuous IV infusion.
Procedure: Radiation Therapy — External Beam Radiotherapy (weeks 1-6), Monday through Friday.

SUMMARY:
The purpose of this study is to test a new treatment of pancreatic cancer that cannot be removed by surgery. This treatment is a Phase I dose escalation research study which will combine one drug at increasing doses with a fixed dose of a second drug and radiation therapy. The drug that will be used at increasing doses is gemcitabine whereas 5-fluorouracil will remain the same for all patients.

DETAILED DESCRIPTION:
* Ultimately we plan to find the maximum tolerated dose of the combination of gemcitabine, 5-fluorouracil and radiation therapy. We also hope to assess the number of people who respond to this therapy and to assess the feasibility of giving intraoperative radiation therapy following gemcitabine, 5-fluorouracil, and external beam radiation therapy.
* A surgical procedure, either laparotomy or laparoscopy, will be required to check the amount of disease before treatment is started.
* All patients will receive the same two chemotherapy drugs and radiation therapy. Both gemcitabine and 5-fluorouracil will begin on the first week of radiation therapy. 5-fluorouracil will be given continuously by intravenous infusion and will continue until the external beam radiation therapy is completed. The gemcitabine will be given (at different doses for each cohort of patients) once per week for seven weeks. Radiation therapy will be given daily for five days for seven weeks. On those days when gemcitabine is given, radiation therapy will be given approximately four hours after the gemcitabine dose.
* Four weeks after completing the radiation therapy and chemotherapy, patients will undergo a scan to check the extent of disease. Following the scan, patients will be considered for a repeat surgical procedure to remove the tumor, if possible. If removal of the tumor is not possible, patients will receive intraoperative radiation therapy.
* After completing the therapy, patients will be seen at least every 3 months for one year. A complete physical exam and CT scan will be done regularly.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of locally unresectable pancreatic adenocarcinoma. Patients with either measurable of evaluable disease are eligible.
* Unresectable, non-metastatic tumors. Unresectable patients include those with local extension of the tumor into adjacent structures and/or nodal metastasis.
* Total bilirubin < 2.0 mg/dl
* AST < 3x ULN
* Serum creatinine < 2.0 mg/dl
* WBC > 3,000/mm3
* Platelets > 100,000/mm3
* ECOG performance status < or = to 2
* Life expectancy of greater than 12 weeks

Exclusion Criteria:

* Evidence of peritoneal seeding by malignancy
* Prior radiation therapy or chemotherapy for pancreatic cancer
* Myocardial infarction in the past 6 months
* Major surgery in past two weeks
* Uncontrolled serious medical or psychiatric illness
* Pregnant or lactating women
* Concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1998-01; Primary Completion 2007-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose of weekly gemcitabine when administered with continuous infusion 5-fluorouracil and external beam radiation. | phase 1

SECONDARY OUTCOMES:
To determine the safety if this regimen | phase 1
to obtain a preliminary assessment of the efficacy of this regimen in this patient population. | phase 1

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Fuchs, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts